CLINICAL TRIAL: NCT03684538
Title: The Efficacy Of Probiotics Versus Zinc Versus Probiotics-Zinc Combination On Acute Diarrhea In Children: A Double Blind Clinical Trial
Brief Title: Efficacy Of Probiotics vs. Zinc vs. Probiotics-Zinc Combination On Acute Diarrhea In Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Mariam Rajab, Pediatrician, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1022018
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Acute Diarrhea
MeSH Terms: interventions — Probiotics; Zinc; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Probiotics (Experimental): Patients in this group will be given the standard of care (initiation of hydration and early refeeding, in addition to the use of antimicrobials in case a pathogen was identified). In addition to that, the patients in this group will receive probiotics (Saccharomyces boulardii) one dose per day.
  Interventions: Other: Probiotics; Other: Standard care
- Group Zinc (Experimental): Patients will be given the standard of care (initiation of hydration and early refeeding, in addition to the use of antimicrobials in case a pathogen was identified). In addition to that, the patients in this group will receive zinc (10 mg for patients less than 6 month and 20 mg for older patients) one dose per day.
  Interventions: Other: Zinc; Other: Standard care
- Group Probiotics & Zinc (Active Comparator): Patients will be given the standard of care (initiation of hydration and early refeeding, in addition to the use of antimicrobials in case a pathogen was identified). In addition to that, the patients in this group will receive a combination of probiotics (Saccharomyces boulardii) with zinc (10 mg for patients less than 6 month and 20 mg for older patients) one dose per day.
  Interventions: Other: Probiotics & Zinc; Other: Standard care

INTERVENTIONS:
Other: Probiotics — Patients will receive probiotics (Saccharomyces boulardii) one dose per day (250 mg)
  Arms: Group Probiotics
Other: Zinc — Patients will receive zinc (10 mg for patients less than 6 month and 20 mg for older patients) one dose per day
  Arms: Group Zinc
Other: Probiotics & Zinc — Patients will receive a combination of probiotics (Saccharomyces boulardii 250 mg) with zinc (10 mg for patients less than 6 month and 20 mg for older patients) one dose per day
  Arms: Group Probiotics & Zinc
Other: Standard care — initiation of hydration and early refeeding, in addition to the use of antimicrobials in case a pathogen was identified

SUMMARY:
Background: Acute diarrhea in children is still a major health burden worldwide despite all efforts that have been made to reduce its incidence and prevalence. Children are more prone for dehydration that is the most common serious complication of acute diarrhea and can be easily avoided. Initiation of rehydration, early refeeding and giving suitable antimicrobial agents when indicated are the cornerstone for management. In addition, studies have emphasized on the role and efficacy of probiotics and zinc supplements on acute diarrhea in children. Indeed, there are a lot of studies on the role of zinc and probiotic in reducing the severity of acute diarrhea, but not many studies have compared effect of using a combination zinc with probiotics to zinc alone and probiotics alone on acute diarrhea.

Objective:To compare the effectiveness of use of probiotics only, zinc only, and combination of zinc with probiotics on the duration and consistency of diarrhea in children presented for acute gastroenteritis.

Methods: A total of 240 patients diagnosed with acute diarrhea will be divided into three groups each of 80 patients. The first group will be managed by addition of probiotics to standard treatment. The second group will be managed by addition of zinc to the standard treatment. The third group will be managed by the addition to a combination of zinc and probiotics to standard treatment. The patients will be followed to compare the effect of the given medication on the duration of diarrhea.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blinded, clinical trial that will be conducted on children presenting with acute diarrhea in Makassed General Hospital.

Patient's level of dehydration will be assessed and a base line of frequency and consistency of diarrhea will be taken from parents'/ caregivers' history and observation. The consistency of stools will be scored according to the "Bristol Stool Chart". Also parents will be asked to sign an informed consent.

A total of 240 eligible patients will be randomized by computer-generated numbers and the sealed envelope technique will be used to divide the patients into three groups.

Group A will be composed of 80 patients. All of them will be given the standard of care (initiation of hydration and early refeeding, in addition to the use of antimicrobials in case a pathogen was identified). In addition to that, the patients in this group will receive probiotics (saccharomyces boulardii) one dose per day.

Group B which will be composed of 80 patients. All of them will be given the standard of care (initiation of hydration and early refeeding, in addition to the use of antimicrobials in case a pathogen was identified). In addition to that, the patients in this group will receive zinc (10 mg for patients less than 6 month and 20 mg for older patients) one dose per day.

Group C which will be composed of 80 patients. All of them will be given the standard of care (initiation of hydration and early refeeding, in addition to the use of antimicrobials in case a pathogen was identified). In addition to that, the patients in this group will receive a combination of probiotics (saccharomyces boulardii) with zinc (10 mg for patients less than 6 month and 20 mg for older patients) one dose per day.

Upon assigning the group (A, B or C), the patient will receive his daily dose of medication in a sealed opaque tiny bag prepared by the nursing staff by adding 5 ml water to the assigned medication which will be unknown to both parent and researcher.

Patients will be assessed on a daily basis. The quality and quantity of diarrhea, as well as hydration status, Po intake and parents satisfaction will be assessed daily until the end of illness, the length of stay for hospitalized patient will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Acute diarrhea
* Patients whose parents signed informed consent
* Patients who have dehydration according to the World Health Organization (WHO) clinical scale

Exclusion Criteria:

* Severe dehydration
* Coexisting severe infection (e.g. sepsis, pneumonia, meningitis)
* Immune deficiency
* Patients whose parents refuse to provide written informed consent
* Patients who do not comply with treatment

Ages: 31 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Diarrhea consistency | Till the end of diarrhea, an average of five days
  consistency of diarrhea scored according to the "Bristol Stool Chart"

SECONDARY OUTCOMES:
Diarrhea duration | Till the end of diarrhea, an average of five days
  duration of diarrhea in days
Hospital stay | Till the end of diarrhea, an average of four days
  Length of hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Mariam AlAbdullah A Rajab, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon

REFERENCES:
- [Derived] Collinson S, Deans A, Padua-Zamora A, Gregorio GV, Li C, Dans LF, Allen SJ. Probiotics for treating acute infectious diarrhoea. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD003048. doi: 10.1002/14651858.CD003048.pub4. PMID 33295643